CLINICAL TRIAL: NCT02391584
Title: XprESS Eustachian Tube Dilation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Entellus Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2909-001
Record Dates: First submitted 2015-03-09; First posted 2015-03-18 (Estimated); Results first posted 2018-11-01 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Eustachian Tube Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- XprESS (Experimental): Balloon dilation of the Eustachian tube
  Interventions: Device: XprESS
- Control (Other): Continued medical management
  Interventions: Other: Control

INTERVENTIONS:
Device: XprESS — Balloon dilation of the Eustachian tube
  Arms: XprESS
Other: Control — Continued medical management
  Other Names: Continued medical management
  Arms: Control

SUMMARY:
Study to assess the safety and efficacy of the XprESS device for transnasal Eustachian tube dilation.

DETAILED DESCRIPTION:
Prospective, multicenter, randomized controlled trial comparing balloon dilation of the Eustachian tube to continued medical management for treatment of persistent Eustachian tube dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Have been diagnosed with symptoms of chronic Eustachian tube dysfunction for no less than 12 months prior to enrollment
* Have an overall ETDQ-7 score ≥3.0
* Have record of failed medical management for Eustachian tube dysfunction

Exclusion Criteria:

* Require concomitant procedures at the time of the study enrollment or procedure
* Have patulous Eustachian tube
* Have ear tubes in place or perforation of the tympanic membrane
* Have evidence of internal carotid artery dehiscence
* Be pregnant at the time of enrollment
* Be currently participating in other drug or device studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-02; Primary Completion 2017-03 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Colorado Sinus Institute, Denver, Colorado
  - Ear Nose Throat and Sinus Clinic, North Platte, Nebraska
  - Donald Guthrie Foundation, Sayre, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Austin Ear Clinic, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Meyer TA, O'Malley EM, Schlosser RJ, Soler ZM, Cai J, Hoy MJ, Slater PW, Cutler JL, Simpson RJ, Clark MJ, Rizk HG, McRackan TR, D'Esposito CF, Nguyen SA. A Randomized Controlled Trial of Balloon Dilation as a Treatment for Persistent Eustachian Tube Dysfunction With 1-Year Follow-Up. Otol Neurotol. 2018 Aug;39(7):894-902. doi: 10.1097/MAO.0000000000001853. PMID 29912819
- [Derived] Swords C, Smith ME, Patel A, Norman G, Llewellyn A, Tysome JR. Balloon dilatation of the Eustachian tube for obstructive Eustachian tube dysfunction in adults. Cochrane Database Syst Rev. 2025 Feb 26;2(2):CD013429. doi: 10.1002/14651858.CD013429.pub2. PMID 40008607

RESULTS

PARTICIPANT FLOW:
Period: Primary Endpoint (6-weeks)
Arm/Group | XprESS | Control
Started | 31 | 29
Completed | 29 | 27
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 1 | 2
Not completed — Missed primary endpoint visit | 1 | 0
Period: 3 Month
Arm/Group | XprESS | Control
Started (Control participants crossed over to balloon dilation or exited the study after the 6-week visit.) | 53 (Includes 30 balloon dilation and 23 crossover participants) | 0 (23 Crossover participants are included in balloon dilation arm for remainder of study visits.)
Completed | 52 | 0
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: 6 Month
Arm/Group | XprESS | Control
Started | 52 | 0
Completed | 51 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: 12 Month (End of Study)
Arm/Group | XprESS | Control
Started | 51 | 0
Completed | 49 | 0
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | XprESS | Control | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (15.4) | 46.6 (15.7) | 49.4 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 31
  Male | 14 | 15 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 28 | 26 | 54
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 29 | 60
Duration of ETD (years) [Mean (Standard Deviation); unit: years] | 12.2 (17.0) | 13.0 (17.3) | 12.6 (17.0)
Baseline mean overall ETDQ-7 score [Mean (Standard Deviation); unit: units on a scale] — The 7-item Eustachian Tube Dysfunction Questionnaire (ETDQ-7) is a validated patient-reported tool measuring ETD symptoms and severity. The 7 items are: pressure in the ears, pain in the ears, a feeling that ears are clogged or underwater, ear symptoms when you have a cold of sinusitis, cracking or popping sounds in the ear, ringing in the ears, and a feeling that your hearing is muffled. Each item is rated from 1 (no problem) to 7 (severe problem) and a mean is calculated for the overall score (range from 1-7). Scores of 1-2 indicate no to mild symptoms, 3-5 moderate, and 6-7 severe symptoms.
  units on a scale | 4.6 (1.1) | 5.0 (0.8) | 4.7 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Overall ETDQ-7 Scores
Description: Comparison of mean change in overall ETDQ-7 scores from baseline to 6 weeks between randomized arms.
  The 7-item Eustachian Tube Dysfunction Questionnaire (ETDQ-7) is a validated patient-reported tool measuring ETD symptoms and severity. The 7 items are: pressure in the ears, pain in the ears, a feeling that your ears are clogged or underwater, ear symptoms when you have a cold of sinusitis, cracking or popping sounds in the ear, ringing in the ears, and a feeling that your hearing is muffled. Each item is rated from 1 (no problem) to 7 (severe problem) and a mean is calculated for the overall score (range from 1-7). Scores of 1-2 indicate no to mild symptoms, 3-5 moderate, and 6-7 severe symptoms.
Time Frame: 6 weeks post procedure (treatment arm) or randomization (control arm)
Population: All randomized participants with completed ETDQ-7 questionnaire at 6-week follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | XprESS | Control
Number analyzed (Participants) | 28 | 27
units on a scale | -2.9 (1.4) | -0.6 (1.0)
Statistical Analysis 1: Comparison: XprESS vs Control; Test type: Superiority; p < 0.0001, t-test, 1 sided — p<0.025 was considered significant

2. Primary Outcome: Complication Rate
Description: Number of subjects who experience serious device- or procedure-related adverse events
Time Frame: Through 6 months post-procedure
Population: All participant's randomized to balloon dilation who underwent the procedure and all control participant's with 6-week follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | XprESS | Control
Number analyzed (Participants) | 30 | 27
Participants | 0 | 0

3. Secondary Outcome: Technical Success Rate
Description: Percent of successful ET dilations per attempted ET dilations
Time Frame: Immediately after procedure
Population: All participants who underwent an attempted unilateral or bilateral balloon dilation of the ET.
Measure: Number; unit: percentage of successful dilations
Units Other Than Participants: ears
Groups:
- All Balloon Dilation Attempts: All Eustachian tubes that underwent an attempted balloon dilation in participants who were randomized to balloon dilation or control participants who crossed over to balloon dilation.
Arm/Group | All Balloon Dilation Attempts
Number analyzed (Participants) | 53
Number analyzed (ears) | 91
percentage of successful dilations | 100

4. Secondary Outcome: Revision Rate
Description: Percent of participants undergoing repeat balloon dilation procedure on an ET that was initially treated with an XprESS device
Time Frame: 12 months
Population: All participants who underwent balloon dilation (randomized and crossover).
Measure: Count of Participants; unit: Participants
Groups:
- All Balloon Dilation Participants: Participants randomized and treated with balloon dilation and control participants who crossed over to balloon dilation.
Arm/Group | All Balloon Dilation Participants
Number analyzed (Participants) | 53
Participants | 0

5. Secondary Outcome: Mean Change in Overall ETDQ-7 Score
Description: Mean change from baseline to 12 months in the overall ETDQ-7 score. The 7-item Eustachian Tube Dysfunction Questionnaire (ETDQ-7) is a validated patient-reported tool measuring ETD symptoms and severity. The 7 items are: pressure in the ears, pain in the ears, a feeling that your ears are clogged or underwater, ear symptoms when you have a cold of sinusitis, cracking or popping sounds in the ear, ringing in the ears, and a feeling that your hearing is muffled. Each item is rated from 1 (no problem) to 7 (severe problem) and a mean is calculated for the overall score (range from 1-7). Scores of 1-2 indicate no to mild symptoms, 3-5 moderate, and 6-7 severe symptoms.
Time Frame: 12 months postdilation
Population: All balloon dilation participants (randomized and crossover) who completed an ETDQ-7 questionnaire at 12-month follow-up.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Balloon Dilation Participants
Number analyzed (Participants) | 49
units on a scale | -2.4 (1.4)
Statistical Analysis 1: Comparison: All Balloon Dilation Participants; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Dunnett's t-test was used for the multiple comparisons with baseline. A p value <0.05 was considered significant

6. Secondary Outcome: Mean Change in Overall ETDQ-7 Score
Description: Mean change from baseline to 6 months in the overall ETDQ-7 score. The 7-item Eustachian Tube Dysfunction Questionnaire (ETDQ-7) is a validated patient-reported tool measuring ETD symptoms and severity. The 7 items are: pressure in the ears, pain in the ears, a feeling that your ears are clogged or underwater, ear symptoms when you have a cold of sinusitis, cracking or popping sounds in the ear, ringing in the ears, and a feeling that your hearing is muffled. Each item is rated from 1 (no problem) to 7 (severe problem) and a mean is calculated for the overall score (range from 1-7). Scores of 1-2 indicate no to mild symptoms, 3-5 moderate, and 6-7 severe symptoms.
Time Frame: 6 months postdilation
Population: All balloon dilation participants (randomized and crossover) who completed an ETDQ-7 questionnaire at 6-month follow-up.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Balloon Dilation Participants
Number analyzed (Participants) | 51
units on a scale | -2.4 (1.4)
Statistical Analysis 1: Comparison: All Balloon Dilation Participants; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Dunnett's t-test was used for the multiple comparisons with baseline. A p value <0.05 was considered significant

7. Secondary Outcome: Mean Change in Overall ETDQ-7 Score
Description: Mean change from baseline to 3 months in the overall ETDQ-7 score. The 7-item Eustachian Tube Dysfunction Questionnaire (ETDQ-7) is a validated patient-reported tool measuring ETD symptoms and severity. The 7 items are: pressure in the ears, pain in the ears, a feeling that your ears are clogged or underwater, ear symptoms when you have a cold of sinusitis, cracking or popping sounds in the ear, ringing in the ears, and a feeling that your hearing is muffled. Each item is rated from 1 (no problem) to 7 (severe problem) and a mean is calculated for the overall score (range from 1-7). Scores of 1-2 indicate no to mild symptoms, 3-5 moderate, and 6-7 severe symptoms.
Time Frame: 3 months postdilation
Population: All balloon dilation participants (randomized and crossover) who completed an ETDQ-7 questionnaire at 3-month follow-up.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Balloon Dilation Participants
Number analyzed (Participants) | 52
units on a scale | -2.5 (1.4)
Statistical Analysis 1: Comparison: All Balloon Dilation Participants; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Dunnett's t-test was used for the multiple comparisons with baseline. A p value <0.05 was considered significant

8. Secondary Outcome: Mean Change in Overall ETDQ-7 Score
Description: Mean change from baseline to 6 weeks in the overall ETDQ-7 score. The 7-item Eustachian Tube Dysfunction Questionnaire (ETDQ-7) is a validated patient-reported tool measuring ETD symptoms and severity. The 7 items are: pressure in the ears, pain in the ears, a feeling that your ears are clogged or underwater, ear symptoms when you have a cold of sinusitis, cracking or popping sounds in the ear, ringing in the ears, and a feeling that your hearing is muffled. Each item is rated from 1 (no problem) to 7 (severe problem) and a mean is calculated for the overall score (range from 1-7). Scores of 1-2 indicate no to mild symptoms, 3-5 moderate, and 6-7 severe symptoms.
Time Frame: 6 weeks postdilation
Population: All balloon dilation participants (randomized and crossover) who completed an ETDQ-7 questionnaire at 6-week follow-up.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Balloon Dilation Participants
Number analyzed (Participants) | 51
units on a scale | -2.5 (1.4)
Statistical Analysis 1: Comparison: All Balloon Dilation Participants; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Dunnett's t-test was used for the multiple comparisons with baseline. A p value <0.05 was considered significant

ADVERSE EVENTS:
Time Frame: 1. 6 weeks between randomized arms (balloon dilation vs control), and 2. 12 months for all participants
Groups:
- XprESS Randomized Arm at 6 Weeks: All participants randomized to balloon dilation and followed through at least the 6-week visit. One randomized balloon dilation participant did not undergo procedure and did not return for the 6-week visit, so this participant is not included in the safety analysis. One other participant did not complete the ETDQ-7 for the primary efficacy endpoint but otherwise completed the rest of the 6-week visit and is therefore included in the safety analysis, resulting in a total XprESS safety population of 30.
- Control Randomized Arm at 6 Weeks: All participants randomized to control and followed through at least the 6-week visit. Two randomized control participants did not return for the 6-week visit, so are not included in the safety analysis resulting in a total control population of 27 for the safety analysis. Control participants who did not crossover were exited from the study after the 6-week visit.
- All Participants Through 12 Months: All participants who were followed through at least the 6-week visit. After the 6-week visit, control participants were either exited or crossed over the balloon dilation.
Arm/Group | XprESS Randomized Arm at 6 Weeks | Control Randomized Arm at 6 Weeks | All Participants Through 12 Months
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/27 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/27 | 0/57
Other Adverse Events (participants affected / at risk) | 2/30 | 1/27 | 13/57
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XprESS Randomized Arm at 6 Weeks (N=30) | Control Randomized Arm at 6 Weeks (N=27) | All Participants Through 12 Months (N=57)
Sinusitis/sinus infection (Infections and infestations) | 2 (2) | 0 (0) | 5 (6)
Ear infection (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 6 (7)
Cold/upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-15): https://cdn.clinicaltrials.gov/large-docs/84/NCT02391584/Prot_SAP_000.pdf